CLINICAL TRIAL: NCT03344822
Title: Place of 68Ga-PSMA-11 PET-CT in the Therapeutic Decision at the End of the Initial Staging for High Risk Prostate Cancer Patients in Comparaison of 18F-Choline PET-CT
Brief Title: Place of 68Ga-PSMA-11 PET-CT in the Therapeutic Decision at the End of the Initial Staging for High Risk Prostate Cancer Patients
Acronym: TePSMAG-68
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSS2016/TePSMAG-68-CLAUDIN/VS
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: 68Ga-PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Each patient will realize a 18F-Choline PET/CT then a 68Ga-PSMA-11 PET/CT
Masking Description: Even if the study has only one arm, the results of both PET imageries will be blind assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA PET-CT (Experimental)
  Interventions: Diagnostic Test: 68Ga-PSMA-11; Diagnostic Test: 18F-Choline PET-CT

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-11 — radioactive tracer for PET-CT (68Ga-PSMA-11)
Diagnostic Test: 18F-Choline PET-CT — radioactive tracer for PET-CT (18F-Choline PET-CT)

SUMMARY:
Several studies have shown a great potential of 68Ga-PSMA PET in high risk prostate cancers patients and a high detection rate than 18F-Choline PET.

The primary aim of this study is to evaluate the difference of management intent, after the inital staging of high risk prostate cancer patients, with 68Ga-PSMA-11 PET-CT results in comparison of 18F-Choline PET-CT results.

ELIGIBILITY:
Inclusion Criteria:

* high risk prostate cancer patients with initial tests : CT, bone scintigraphy and 18F-Choline

Exclusion Criteria:

* contraindication of 68Ga-PSMA PET-CT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of modification of management intent | 1 month
  modification of management intent after 68Ga-PSMA PET-CT and 18F-Choline PET-CT

CONTACTS AND LOCATIONS:
Locations (1):
- Central hospital Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No